CLINICAL TRIAL: NCT01791049
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose (SAD) Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TD-1607, a Glycopeptide-Cephalosporin Heterodimer Gram-Positive Antibiotic, in Healthy Subjects
Brief Title: TD-1607 SAD Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 0098
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Serious Infections Due to Known or Suspected Gram-positive Pathogens
Keywords: Gram-positive; Infections; Bacterial infections
MeSH Terms: conditions — Infections; Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Single escalating doses of TD-1607, administered intravenously
  Interventions: Drug: TD-1607
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-1607
  Arms: Active
Drug: Placebo
  Arms: Placebo

SUMMARY:
TD-1607, administered intravenously as single doses, will be investigated in healthy subjects to assess its tolerability, safety, and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy nonsmoking male or a female of non-child bearing potential and 18 to 50 years old, inclusive, at Screening. Females are considered to be of non-childbearing potential if they have had a hysterectomy or tubal ligation or are postmenopausal (amenorrheic for at least 2 years) with a follicle-stimulating hormone (FSH) level >20 IU/L.
* Subject has a body mass index (BMI) of 19 to 30 kg/m2, inclusive, and weighs at least 50 kg

Exclusion Criteria:

* Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic seasonal allergies at time of dosing), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
* Subject has a history of allergies or hypersensitivities to glycopeptide (e.g., vancomycin), penicillin, or cephalosporin antibiotics.
* Subject has participated in another clinical trial of an investigational drug (or medical device) within 60 days (or 5 half-lives, whichever is longer) prior to Screening or is currently participating in another trial of an investigational drug (or medical device).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 11 days
  Adverse events, laboratory abnormalities, ECGs, and vital sign measurements.

SECONDARY OUTCOMES:
Pharmacokinetics | 96 hours
  Cmax, Tmax, AUC0-t, AUC0-24, AUCinf, CL, Vdss, t1/2, amount excreted in urine (Ae), fraction eliminated in urine (fe), and CLr.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- PPD Phase 1, Austin, Texas, United States